CLINICAL TRIAL: NCT04729283
Title: Prospective Comparative Multicentric Study, Assess the Quality of Life and Functionnal Results After Sigmoidectomy for Diverticulitis and Cancer
Brief Title: Comparison of Quality of Life and Functionnal Resultats After Sigmodectomy Between Diverticulitis and Cancer
Acronym: SIG-QOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0015
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Sigmoid Cancer; Sigmoid Diverticulosis
Keywords: LARS score; Sigmoidectomy; Sigmoid cancer; Diverticulitis; Functional results
MeSH Terms: conditions — Sigmoid Neoplasms; Diverticulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sigmoidectomy for sigmoid cancer: Sigmoid resection surgery for patients who suffer from sigmoid cancer
  Interventions: Procedure: Sigmoidectomy
- Sigmoidectomy for diverticulitis: Sigmoid resection surgery for patients who suffer from symptomatic diverticulitis
  Interventions: Procedure: Sigmoidectomy

INTERVENTIONS:
Procedure: Sigmoidectomy — The sigmoid resection surgery, realized by laparoscopy or laparotomy, with anastomosis.

SUMMARY:
The aim of this present study is to compare functional results and quality of life after sigmoidectomy for diverticulitis and sigmoid cancer.

DETAILED DESCRIPTION:
Rectal resection surgery can lead to numerous complications in term of gastrointestinal results with onset of fecal incontinence or in contrast constipation, and in term of genitourinary results with occurrence of dysuria, erectile dysfunction, or vaginal dryness. The low anterior resection syndrome is defined by the occurrence after rectal resection, of gastrointestinal symptoms like fecal incontinence or stool evacuation difficulties, which affect quality of life, despite conservation of anal sphincter. This syndrome is now well known and used in many countries.

However, there is a lack of data concerning gastrointestinal functional results after sigmoid surgery whether it is for cancer or diverticulitis. Some studies highlighted symptoms persistence in many patients after sigmoidectomy. Lately, the LARS score was used after sigmoidectomy for cancer. This study reveals symptoms of low anterior resection syndrome for 41 % of patients. The correlation between rectal resection and sigmoidectomy could be explain by the resection of the upper part of rectum in case of sigmoidectomy.

The issue of genito-urinary disorders after sigmoidectomy are poorly researched. Previous studies demonstrate a higher risk of erectile disorders after pelvic surgery and especially for cancer.

Currently, there is a lack of data on functional results and quality of life for patients who are going into sigmoid surgery, whether for cancer or diverticulitis. The aim of this longitudinal study is to compare digestive functional outcome, genitourinary outcomes and quality of life in patients who undergo sigmoid resection for diverticulitis and cancer.

ELIGIBILITY:
Inclusion Criteria :

* Adults
* Patients who undergo sigmoidectomy with end to end anastomosis for sigmoid cancer and symptomatic diverticulitis
* Preservation of the left colic angle for upper surgical resection
* Lower surgical resection located < 5cm to the recto-sigmoid junction

Exclusion Criteria :

* Minors
* Adults under guardianship
* Protected persons
* Patients who undergo sigmoidectomy without anastomosis (ileostomy or Hartmann surgery)
* Patients who undergo surgery in emergency
* Cancer of recto-sigmoid junction
* Patients who undergo secondarily a stoma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffered from sigmoid cancer or symptomatic diverticulitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
LARS score | At the visit of preoperative
  To measure incontinence troubles after low anterior resection. The score is from 0 to 42. The higher the score, the worst the incontinence.
LARS score | At the visit of one month
  To measure incontinence troubles after low anterior resection. The score is from 0 to 42. The higher the score, the worst the incontinence.
LARS score | At the visit of three months
  To measure incontinence troubles after low anterior resection. The score is from 0 to 42. The higher the score, the worst the incontinence.
LARS score | At the visit of six months
  To measure incontinence troubles after low anterior resection. The score is from 0 to 42. The higher the score, the worst the incontinence.
LARS score | At the visit of twelve months
  To measure incontinence troubles after low anterior resection. The score is from 0 to 42. The higher the score, the worst the incontinence.

SECONDARY OUTCOMES:
Bristol stool chart | At the visit of preoperative
  A scale to classify the form of the stools in seven category which indicate constipation or diarrhea in function of the type.
  Types 1 and 2 indicate constipation, types 3 and 4 are normal stools, type 5, 6 and 7 indicate diarrhea.
Bristol stool chart | At the visit of one month
  A scale to classify the form of the stools in seven category which indicate constipation or diarrhea in function of the type.
  Types 1 and 2 indicate constipation, types 3 and 4 are normal stools, type 5, 6 and 7 indicate diarrhea.
Bristol stool chart | At the visit of three months
  A scale to classify the form of the stools in seven category which indicate constipation or diarrhea in function of the type.
  Types 1 and 2 indicate constipation, types 3 and 4 are normal stools, type 5, 6 and 7 indicate diarrhea.
Bristol stool chart | At the visit of six months
  A scale to classify the form of the stools in seven category which indicate constipation or diarrhea in function of the type.
  Types 1 and 2 indicate constipation, types 3 and 4 are normal stools, type 5, 6 and 7 indicate diarrhea.
Bristol stool chart | At the visit of twelve months
  A scale to classify the form of the stools in seven category which indicate constipation or diarrhea in function of the type.
  Types 1 and 2 indicate constipation, types 3 and 4 are normal stools, type 5, 6 and 7 indicate diarrhea.
GIQLI | At the visit of preoperative
  Quality of life related to gastrointestinal symptoms. Score from 0 to 144. The higher the score, the better the quality of life.
GIQLI | At the visit of one month
  Quality of life related to gastrointestinal symptoms. Score from 0 to 144. The higher the score, the better the quality of life.
GIQLI | At the visit of three months
  Quality of life related to gastrointestinal symptoms. Score from 0 to 144. The higher the score, the better the quality of life.
GIQLI | At the visit of six months
  Quality of life related to gastrointestinal symptoms. Score from 0 to 144. The higher the score, the better the quality of life.
GIQLI | At the visit of twelve months
  Quality of life related to gastrointestinal symptoms. Score from 0 to 144. The higher the score, the better the quality of life.
SF-36 | At the visit of preoperative
  General quality of life score. Described with 8 scaled scores, which are : vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, social role functioning, mental health.
  Each scale score is from 0 to 100. The higher the score the less disability.
SF-36 | At the visit of one month
  General quality of life score. Described with 8 scaled scores, which are : vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, social role functioning, mental health.
  Each scale score is from 0 to 100. The higher the score the less disability.
SF-36 | At the visit of three months
  General quality of life score. Described with 8 scaled scores, which are : vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, social role functioning, mental health.
  Each scale score is from 0 to 100. The higher the score the less disability.
SF-36 | At the visit of six months
  General quality of life score. Described with 8 scaled scores, which are : vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, social role functioning, mental health.
  Each scale score is from 0 to 100. The higher the score the less disability.
SF-36 | At the visit of twelve months
  General quality of life score. Described with 8 scaled scores, which are : vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, social role functioning, mental health.
  Each scale score is from 0 to 100. The higher the score the less disability.
FSFI | At the visit of preoperative
  Measure of sexual functioning in women. Score from 0 to 95. The higher the score, the better the sexual function.
FSFI | At the visit of one month
  Measure of sexual functioning in women. Score from 0 to 95. The higher the score, the better the sexual function.
FSFI | At the visit of three months
  Measure of sexual functioning in women. Score from 0 to 95. The higher the score, the better the sexual function.
FSFI | At the visit of six months
  Measure of sexual functioning in women. Score from 0 to 95. The higher the score, the better the sexual function.
FSFI | At the visit of twelve months
  Measure of sexual functioning in women. Score from 0 to 95. The higher the score, the better the sexual function.
ICIQ-FLUTS | At the visit of preoperative
  Questionary for evaluating female lower urinary tract symptoms and impact on quality of life.
  Score from 0 to 48. The higher the score, the worst the urinary continence.
ICIQ-FLUTS | At the visit of one month
  Questionary for evaluating female lower urinary tract symptoms and impact on quality of life.
  Score from 0 to 48. The higher the score, the worst the urinary continence.
ICIQ-FLUTS | At the visit of three months
  Questionary for evaluating female lower urinary tract symptoms and impact on quality of life.
  Score from 0 to 48. The higher the score, the worst the urinary continence.
ICIQ-FLUTS | At the visit of six months
  Questionary for evaluating female lower urinary tract symptoms and impact on quality of life.
  Score from 0 to 48. The higher the score, the worst the urinary continence.
ICIQ-FLUTS | At the visit of twelve months
  Questionary for evaluating female lower urinary tract symptoms and impact on quality of life.
  Score from 0 to 48. The higher the score, the worst the urinary continence.
IPSS | At the visit of preoperative
  Questionary to screen and manage symptoms of benign prostatic hyperplasia. Score from 0 to 35. The higher the score, the worst the urinary function.
IPSS | At the visit of one month
  Questionary to screen and manage symptoms of benign prostatic hyperplasia. Score from 0 to 35. The higher the score, the worst the urinary function.
IPSS | At the visit of three months
  Questionary to screen and manage symptoms of benign prostatic hyperplasia. Score from 0 to 35. The higher the score, the worst the urinary function.
IPSS | At the visit of six months
  Questionary to screen and manage symptoms of benign prostatic hyperplasia. Score from 0 to 35. The higher the score, the worst the urinary function.
IPSS | At the visit of twelve months
  Questionary to screen and manage symptoms of benign prostatic hyperplasia. Score from 0 to 35. The higher the score, the worst the urinary function.
IIEF5 | At the visit of preoperative
  Questionary about erection problems on patient's sex life. Score from 1 to 25. The higher the score, the better the sexual function.
IIEF5 | At the visit of one month
  Questionary about erection problems on patient's sex life. Score from 1 to 25. The higher the score, the better the sexual function.
IIEF5 | At the visit of three months
  Questionary about erection problems on patient's sex life. Score from 1 to 25. The higher the score, the better the sexual function.
IIEF5 | At the visit of six months
  Questionary about erection problems on patient's sex life. Score from 1 to 25. The higher the score, the better the sexual function.
IIEF5 | At the visit of twelve months
  Questionary about erection problems on patient's sex life. Score from 1 to 25. The higher the score, the better the sexual function.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Caen University Hospital, Caen, Calvados
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Angers University Hospital, Angers, Maine-et-Loire
  - Vendée Departmental Hospital, La Roche-sur-Yon, Vendée

IPD SHARING:
Plan to Share IPD: No